CLINICAL TRIAL: NCT00084565
Title: Phase II Study of the Activity of Weekly Paclitaxel, Topotecan Plus Oral Estramustine Phosphate in Metastatic Hormone-Refractory Prostate Carcinoma
Brief Title: Paclitaxel, Topotecan, and Estramustine in Treating Patients With Metastatic Hormone-Refractory Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never activated at Fox Chase Cancer Center.
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: FCCC-03035; CDR0000365459 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estramustine; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: estramustine phosphate sodium
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, topotecan, and estramustine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one chemotherapy drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel, topotecan, and estramustine together works in treating patients with metastatic hormone therapy-refractory prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with metastatic hormone-refractory prostate cancer treated with paclitaxel, topotecan, and estramustine.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.

Secondary

* Determine the frequency and number of circulating tumor cells in patients before and after treatment with this regimen and at disease progression.
* Determine the microtubule morphology, β-tubulin isotype pattern, apoptotic markers, and metaphase chromosome alignment in circulating tumor cells in patients before and after treatment with this regimen and at disease progression.

OUTLINE: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15; topotecan IV over 30 minutes on days 2, 9, and 16; and oral estramustine twice daily on days 1 and 2 of course 1 and on days 0-2, 7-9, and 14-16 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 18-38 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate gland

  * Progressive metastatic disease (e.g., bone, pelvic mass, lymph node, liver or lung metastases)
  * Radiologic evidence of hydronephrosis alone dose not constitute metastatic disease
* Failed prior primary hormonal therapy (e.g., estrogen therapy, luteinizing hormone-releasing hormone blocker and flutamide) or bilateral orchiectomy

  * Patients previously treated with flutamide or bicalutamide must have evidence of disease progression i.e., increasing Prostate-Specific Antigen (PSA)
* PSA level ≥ 10 ng/mL if bone metastases only are present (i.e., lacking measurable soft tissue disease)
* No elevated serum acid phosphatase or PSA level as the only evidence of disease
* No carcinomatous meningitis or brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* White Blood Cell (WBC) ≥ 4,000/mm^3 OR
* Granulocyte count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Serum Glutamic-Oxaloacetic Transaminase(SGOT) and Serum Glutamic-Pyruvic Transaminase (SGPT) ≤ 2 times normal
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine ≤ 2.0 mg/dL OR
* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* History of deep venous thrombosis allowed provided patients are maintained on therapeutic anticoagulation therapy
* No active angina pectoris
* No New York Heart Association class II-IV heart disease
* No myocardial infarction within the past 6 months
* No thrombosis within the past 3 months

Other

* Fertile patients must use effective contraception during and for 3 months after study participation
* No active infection
* No other concurrent serious medical illness that would preclude study participation
* No other malignancy within the past 3 years except curatively treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior flutamide
* At least 8 weeks since prior bicalutamide

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium

Surgery

* See Disease Characteristics

Other

* Recovered from all prior therapy
* No prior cytotoxic therapy for prostate cancer
* No concurrent milk, milk products, antacids, calcium-containing drugs, or food during estramustine administration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-11; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Hudes, MD, Principal Investigator — Fox Chase Cancer Center